CLINICAL TRIAL: NCT01684202
Title: A Multicenter, Open-label, Dose-finding Trial of OPC-41061 to Investigate Efficacy, Pharmacokinetics, Pharmacodynamics, and Safety in Patients With Carcinomatous Edema (Phase 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-12-001; JapicCTI-121957 (Other: JAPIC)
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Carcinomatous Edema
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-41061 (Experimental)
  Interventions: Drug: OPC-41061

INTERVENTIONS:
Drug: OPC-41061 — orally administered at 3.75, 7.5, 15, or 30 mg once daily after breakfast for up to 11 days.

SUMMARY:
OPC-41061 will be administered to patients with volume overload associated with cancer, first by dose-escalation and subsequently for 6 consecutive days at the fixed dose at which urine volume is increased to investigate efficacy, pharmacokinetics, pharmacodynamic effects, and safety and to determine the effective initial and maintenance doses of OPC-41061.

ELIGIBILITY:
Inclusion Criteria:

* Subjects judged as having cancer by biopsy or cytology
* Subjects with carcinomatous ascites
* Male or female subjects between the ages of 20 and 80, inclusive (at time of informed consent)
* Subjects with survival expectancy of at least 3 months and an Eastern Cooperative Oncology Group (ECOG) Performance Status score (PS score) of 0 to 2
* Subjects who are inpatients or who can be admitted to the trial site for the duration of the trial
* Subjects who, together with their partner, are able to practice one of the specified contraceptive methods until 4 weeks after final trial drug administration
* Subjects capable of giving informed consent to participate in the trial of their own free will prior to start of the trial.

Exclusion Criteria:

* Subjects with any of the following complications or symptoms:

  * Deep vein thrombosis
  * Intestinal obstruction or intestinal edema with symptoms similar to intestinal obstruction
  * Hepatic cirrhosis
  * Anuria
  * Urination impaired due to urinary tract stricture, urinary calculus, tumor in urinary tract, or other cause
  * Continuing symptoms of diarrhea or vomiting
  * Infection requiring systemic treatment
* Subjects with any of the following medical histories:

  * History of cerebrovascular disorder or coronary disease within 4 weeks prior to start of the pre-observation period
  * History of hypersensitivity or idiosyncratic reaction to benzazepine derivatives such as mozavaptan hydrochloride or benazepril hydrochloride
  * History of gastrectomy or enterectomy to an extent affecting absorption of oral medication
* Subjects with any of the following abnormal laboratory values:

Platelet count of < 75,000/mm3, hemoglobin of < 8.0 g/dL, neutrophil count of < 1,000/mm3, total bilirubin of > 4.0 g/dL, serum creatinine of > 3.0 mg/dL, serum sodium of > 147 mEq/L, or serum potassium of > 5.5 mEq/L

* Subjects who have used albumin products (agents for treating hypoalbuminemia) or blood products containing albumins within 1 week prior to start of the pre-observation period, or after start of the pre-observation period
* Subjects who have received any investigational drug within 4 weeks prior to start of the pre-observation period
* Subjects who have previously received OPC-41061
* Subjects who have received surgical treatment or radiation therapy for cancer within 4 weeks prior to start of the pre-observation period
* Subjects for whom the investigator or subinvestigator judges that it would be difficult to evaluate the efficacy and safety of OPC-41061 due to the effects of ongoing chemotherapy or other therapies for cancer (eg, improvement of carcinomatous ascites or development of edema due to adverse events related to therapeutic interventions other than OPC-41061)
* Subjects who are unable to sense thirst or who have difficulty with fluid or food intake
* Subjects who are unable to take oral medication
* Female subjects who are pregnant, possibly pregnant, or nursing, or who plan to become pregnant during the trial period Subjects otherwise judged by the investigator or subinvestigator to be inappropriate for inclusion in the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Hahimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kansai Region, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- OPC-41061 3.75 mg; OPC-41061 7.5 mg; OPC-41061 15 mg; OPC-41061 30 mg: Orally administered at 3.75, 7.5, 15, or 30 mg once daily after breakfast for up to 11 days, first in a dose-escalation manner until daily urine volume increased by 500 mL or more from that at the end of the pretreatment observation period, and then for 6 consecutive days at the fixed dose at which that increase in daily urine volume was achieved. Each Arm/Group Title indicated the final dose.
Period: Dose-escalation Period
Arm/Group | OPC-41061 3.75 mg | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg
Started | 15 | 8 | 9 | 11
Completed | 14 | 7 | 9 | 11
Not Completed | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | OPC-41061 3.75 mg | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg
Started | 14 | 7 | 9 | 11
Completed | 13 | 4 | 8 | 10
Not Completed | 1 | 3 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: all subjects who had been administered the investigational medicinal product (IMP) at least once and from whom data for efficacy endpoints were obtained after the start of IMP administration.
Groups:
- OPC-41061 3.75 mg: Orally administered at 3.75 mg once daily in maintenance period.
- OPC-41061 7.5 mg: Orally administered at 7.5 mg once daily in maintenance period.
- OPC-41061 15 mg: Orally administered at 15 mg once daily in maintenance period.
- OPC-41061 30 mg: Orally administered at 30 mg once daily in maintenance period.
- Total: Total of all reporting groups
Arm/Group | OPC-41061 3.75 mg | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg | Total
Number analyzed (Participants) | 13 | 7 | 9 | 11 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.9) | 66.1 (8.5) | 62.2 (7.6) | 69.5 (7.9) | 65.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 7 | 7 | 24
  Male | 7 | 3 | 2 | 4 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 13 | 7 | 9 | 11 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 13 | 7 | 9 | 11 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight From Baseline at Final IMP Administration
Description: Body weight was measured in 100-g units before breakfast and after subjects had urinated at least once, taking care to minimize fluctuations due to defecation or clothing.
Time Frame: Baseline, at the final IMP administration (shortest:7days longest:12days)
Population: Full analysis set: all subjects who had been administered the IMP at least once and from whom data for efficacy endpoints were obtained after the start of IMP administration.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | OPC-41061 3.75 mg | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg
Number analyzed (Participants) | 13 | 7 | 9 | 11
Kg | -0.69 (2.51) | -0.34 (1.99) | -1.13 (1.62) | 0.70 (1.56)

2. Primary Outcome: Change in Ascites Volume From Baseline Measured by Computer Tomography (CT) at Final IMP Administration
Time Frame: Baseline, at the final IMP administration (shortest:7days longest:12days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | OPC-41061 3.75 mg | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg
Number analyzed (Participants) | 11 | 4 | 8 | 10
mL | -77.20 (982.19) | 513.97 (653.30) | 153.72 (993.63) | 539.93 (659.36)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the start of IMP administration up to 10 days after the final IMP administration.
Description: Safety analysis set: all subjects who had been administered the IMP at least once.
Arm/Group | OPC-41061 3.75 mg | OPC-41061 7.5 mg | OPC-41061 15 mg | OPC-41061 30 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/8 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/8 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 8/15 | 6/8 | 8/9 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-41061 3.75 mg (N=15) | OPC-41061 7.5 mg (N=8) | OPC-41061 15 mg (N=9) | OPC-41061 30 mg (N=11)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-41061 3.75 mg (N=15) | OPC-41061 7.5 mg (N=8) | OPC-41061 15 mg (N=9) | OPC-41061 30 mg (N=11)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 2 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Thirst (General disorders) | 1 | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Stitch abscess (Infections and infestations) | 0 | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 0
Blood osmolarity increased (Investigations) | 1 | 1 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram T wave peaked (Investigations) | 0 | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 1 | 0
Urine ketone body (Investigations) | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No